CLINICAL TRIAL: NCT00399295
Title: An Open-Label Evaluation of the Independent Effect of Coadministration of a High Fat Meal and Naltrexone Blockade on the Pharmacokinetic Profile of Dilaudid OROS (Hydromorphone HCL) 16 mg
Brief Title: An Open-Label Evaluation of the Independent Effects of Coadministration of a High-Fat Meal and Naltrexone Blockade on the Pharmacokinetic Profile of Dilaudid OROS (Hydromorphone HCI) 16mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR011608
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Analgesia
Keywords: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Naltrexone; Narcotic Antagonists

INTERVENTIONS:
Drug: Hydromorphone HCL 16mg; Dilaudid SR 16mg; Naltrexone (opioid antagonist) 50mg.

SUMMARY:
The purpose of this study was to compare the pharmacokinetic (the way a drug enters and leaves the blood and tissues over time) profile of Dilaudid OROS 16mg (Dilaudid Slow Release; hydromorphone HCL) administered under fasting conditions, following a high-fat breakfast meal. The study also examined the effect of naltrexone blockade on the pharmacokinetic profile of Dilaudid SR.

DETAILED DESCRIPTION:
This was a randomized (patients are assigned different treatments based on chance), open-label, three-way crossover study, performed in normal, healthy adults. Each patient received orally administered treatments (a different treatment during each dosing phase): Treatment A: single dose of Dilaudid SR 16 mg administered under fasting conditions without the naltrexone block;Treatment B: single dose of Dilaudid SR 16 mg administered under fed conditions without the naltrexone block, Treatment C: single dose of Dilaudid SR 16 mg administered under fasting conditions with naltrexone HCL 50mg block (3 oral doses of 50mg each administered 12 hours prior to , at the time of, and 12 hours after Dilaudid SR 16mg administration). There was a 7-day washout period between dosing phases.

Venous blood sampling times were 0 (prior to dosing),2,4,6,8,10,12,16,20,24,30,36,42,and 48 hours after each Dilaudid SR administration. LC/MS/MS (Liquid Chromatography/Mass Spectroscopy/Mass Spectroscopy)techniques were employed for the analysis of plasma for hydromorphone concentration. Each patient randomly received orally-administered treatments of single dose of Dilaudid SR 16mg; under fasting conditions without the naltrexone block; under fed conditions without naltrexone block; under fasting conditions with naltrexone 50mg block (3 oral doses of 50mg naltrexone HCL each administered 12 hours prior to, at the time of, and 12 hours after hydromorphone administration); 7-day washout period between dosing phases.

ELIGIBILITY:
Inclusion Criteria:

* Patients were non-smoking, healthy volunteers with body weights between 135 and 220 pounds and within + - 10% of their recommended weight range for their height and body frame according to the 1984 Metropolitan Height and Weight Tables
* A negative baseline urine drug screen for cannabinoids, opiates, cocaine, ethanol and barbiturates.

Exclusion Criteria:

* Patients intolerant of or hypersensitive to hydromorphone or naltrexone
* Patients with any gastrointestinal disorder that may affect the absorption of orally administered drugs
* Patient with depressed respiratory function
* Patient with impaired renal or hepatic function
* Patients with dependence to opiates
* Pregnant or breast feeding
* Female Patients of childbearing potential must have a negative pregnancy test each week prior to administration of study drug and required to be following a medically recognized contraceptive program prior to and during the study.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Study Completion 1997-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoints for the statistical evaluations of the study drug were: Area Under the Concentration-Time Curve from 0 to Infinity and Peak Plasma Concentration.

SECONDARY OUTCOMES:
Secondary endpoints were the parameters for the study drug: Area Under the Concentration-Time Curve from 0 to Time t, Time to Peak Plasma Concentration and Terminal Half Life).

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- [Derived] Sathyan G, Xu E, Thipphawong J, Gupta SK. Pharmacokinetic profile of a 24-hour controlled-release OROS formulation of hydromorphone in the presence and absence of food. BMC Clin Pharmacol. 2007 Feb 2;7:2. doi: 10.1186/1472-6904-7-2. PMID 17270055